CLINICAL TRIAL: NCT00983333
Title: Beta Test of the Time to Talk CARDIO (Creating a Real Dialogue In the Office) Web-based Tool for Improving Communication Between Patients and Health Care Professionals
Brief Title: Initial Test of the Time to Talk CARDIO (Creating a Real Dialogue In the Office) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cliff Coleman, Assistant Professor of Family Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OHSU00005635
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Disease; Cardiovascular Risk Factors
Keywords: Health communication; Health literacy; Patient; Health Care Professional; Satisfaction
MeSH Terms: conditions — Cardiovascular Diseases; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Web-based communication tool for health care professionals (Experimental)
  Interventions: Device: Time to Talk CARDIO website
- Web-based communication training tool for patients (Experimental)
  Interventions: Device: Time to Talk CARDIO website
- Usual care for patient participants (No Intervention)

INTERVENTIONS:
Device: Time to Talk CARDIO website — This interactive web-based training device involves the completion of a brief survey regarding communication experiences between patients and health care professionals. The pattern of responses to the survey generates a personalized set of short instructional videos which demonstrate effective communication skills.
  Arms: Web-based communication tool for health care professionals; Web-based communication training tool for patients

SUMMARY:
This research focuses on communication practices between patients and health care professionals, like nurses, doctors, or physician assistants. The goal is to help improve communication about heart health issues.

This pilot (or Beta) study is designed to test our ability to recruit an appropriate sample of participants, and determine our ability to deliver and evaluate the effects of a web-based intervention. The investigators hypothesize that exposure to the intervention will result in measurable changes in self-reported knowledge, attitudes and behavior regarding communication between patients and health care professionals.

Participants in this research study are being recruited from the people who currently receive care at the Richmond Family Health Center of the Oregon Health & Science University. People who participate in this study will be between 55 and 70 years old, speak English as their preferred language, and have one of several possible diagnoses related to heart health. These could include, for example, hypertension, diabetes, asthma, or obesity.

Additionally, the investigators are recruiting a small number of health care professionals from the Richmond Family Health Center. Their participation will be similar to but separate from the participation of patients.

All participants will take two web-based surveys. Some participants will use a web-based tool that hopes to help improve communication between health care professionals and patients.

The surveys contain questions that explore the knowledge, attitudes, and behaviors of participants related to heart health and communication between health care professionals and patients.

Data analysis will focus upon identifying any changes that occurred in knowledge, attitudes, or behaviors with respect to health communication after using the web-based tool, as well as learning about what influences the quality and nature of communication between health care professionals and the patients they serve.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-70 years
* English is preferred language
* Has one or more chronic cardiovascular-related diagnosis or risk factor
* Has an appointment with Primary Care provider within 2 weeks of enrollment

Exclusion Criteria:

* Inadequate vision or hearing to complete on-line assessment

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Interpersonal communication knowledge, attitudes and behaviors exhibeted by patients and health care professionals during a patient-provider office visit | 2 weeks

SECONDARY OUTCOMES:
Patient and health care professional satisfaction with communication | 2 weeks
Change in patient average blood pressure | 6 months
Change in serum hemoglobin A1c value among patients with diabetes | 6 months
change in average appointment length for health care professionals | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A Coleman, MD, MPH, Principal Investigator — Oregon Health and Science University; Andrew F Pleasant, Ph.D., Study Director — Canyon Ranch Institute
Locations (1):
- Richmond Family Health Center at Oregon Health & Science University, Portland, Oregon, United States